CLINICAL TRIAL: NCT01696721
Title: Proton and Photon Consortium Registry (PPCR): A Multi Center Registry of Pediatric Patients Treated With Radiation Therapy
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Torunn Yock, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 12-103
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Patients Treated With Radiation Therapy
Keywords: Proton Therapy; Pediatrics; Radiation Oncology; Photon Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Patients Treated with Protons: Proton Radiation Therapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
In previous studies, Proton Beam Radiation Therapy (PBRT) has been found to show better results in treating patients with cancer, both because there is better control of where in the body the radiation is directed and because it is associated with less severe long term side effects. However, there is limited published data demonstrating these results. The goal of the Proton and Photon Consortium Registry (PPCR) is to enroll children treated with radiation in order to describe the population that currently receives radiation and better compare the short-term and long-term benefits of different types of radiotherapy. The data collected from this study will help facilitate research on radiation therapy and allow for collaborative research. The PPCR will collect demographic and clinical data that many centers that deliver radiation therapy already collect in routine operations.

DETAILED DESCRIPTION:
Once you are enrolled in the study, you will receive treatment, evaluations and follow up care for your type of cancer as determined by your treating physician according to clinical judgment and standard of care for your clinic. All treatments that you receive will be recorded, including all surgeries and chemotherapy given before or after PBRT. Treatment outcomes, like how you respond to treatment, side effects, and progression of your cancer will be collected as the information becomes available. A study coordinator or research nurse at your clinic will perform a chart review annually to update your status in the database. The study doctor will request any new data within the past year from you or your doctor.

We will be collecting the following data for the Registry:

At Screening: The following data will be collected from the time of diagnosis and initial staging:

* Patient demographics, date of birth, gender, race, zip code and insurance status
* Date of diagnosis
* Histologic or clinical diagnosis and staging relevant to diagnosis
* Imaging studies obtained and tumor measurements
* Lab evaluations which include routine blood tests, hormone levels, and any relevant lab results needed to assess you and baseline and follow-up visits
* Referring physician contact information

Treatment Data Collection: The following data regarding treatment will be collected:

* Treatments received before radiation therapy, including surgery, chemotherapy, dates and numbers of cycles, results of chemotherapy if available
* Dates and doses of radiation treatment
* Side effects observed
* Any treatments you received at the same time as proton radiation therapy

Follow-up Data Collection: The following data will be collected either as it comes in or annually following completion of your radiation therapy treatment:

* Disease and survival status
* Hospitalization, surgeries or other procedures
* New diagnoses of medical conditions
* Any lab results, including x-rays
* Medications you are taking
* Late side effects such as hearing loss, hormonal issues, any cardiac issues
* Development of any new types of cancers
* Dates of treatment after radiation therapy
* If you discontinued radiation therapy
* Laboratory/physician/dental or psychological evaluations
* Use of special services in school (IEP, FM hearing system, one on one tutor, special education) We would like to keep track of your medical condition for the rest of your life. We would like to do this by contacting you or your doctor once a year to see how you are doing. Keeping in touch with you and checking on your condition helps determine the long-term outcomes of individuals treated with proton beam radiation therapy.

In addition to research personnel at MGH, there are others that may have access to the data collected. This includes:

* Other research doctors and medical centers participating in this research, if applicable
* Outside individuals or entities that have a need to access this information to perform functions relating to the conduct of this research. For instance copies of your imaging studies and treatment plan will be stored at MIMcloud. MIMcloud is a service offered through MIM Software Inc, a privately held company, that provides diagnostic imaging data management services.

ELIGIBILITY:
Eligibility Criteria:

1. Patients treated with radiation therapy at one of the participating centers
2. Age < 22 at time of treatment start.
3. Patients may be enrolled regardless of previous local or systemic treatments received prior to enrollment in the PPCR.
4. Patients may be enrolled regardless of other current local or systemic treatments or disease extent.
5. Patients may be enrolled on the PPCR concurrently with another study or clinical trial.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients age <22 treated with radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Establish Registry | 2 years
  Establish a registry of pediatric patients treated with proton radiation therapy in the United States

SECONDARY OUTCOMES:
Describe patterns of care | 2 years
  Describe the patterns of care for pediatric patients receiving proton radiation therapy
Describe patterns of follow-up | 2 years
  Describe the patterns of follow-up at proton facilities where patients are often referred from a significant distance and from centers of excellence
Describe acute and late effects | 2 years
  Describe the acute and late effects in the children treated with proton radiotherapy
Establish a cohort of photon-treated patients | 2 years
  Establish a control group of patients treated with photon radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Torunn I Yock, MD, Principal Investigator — Massachusetts General Hospital
Locations (26):
- United States (24):
  - Stanford University, Palo Alto, California
  - California Protons Cancer Therapy Center, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Florida Health Proton Therapy Institute, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - ProCure Proton Therapy Center- New Jersey, Somerset, New Jersey
  - New York Proton Center, New York, New York
  - State University of New York Upstate Medical Center, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Cincinnati Children's Proton Therapy Center, Liberty Township, Ohio
  - Oklahoma Proton Center, Oklahoma City, Oklahoma
  - ProCure Proton Therapy Center- Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania - Roberts Proton Therapy Center, Philadelphia, Pennsylvania
  - Provision Center for Proton Therapy, Knoxville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Center for Proton Therapy, Irving, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington- Seattle Cancer Care Alliance, Seattle, Washington
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- University Health Network - Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Krisch JM, Ermoian RP, Indelicato DJ, Lee JY, Perentesis JP, Perkins SM, Laack NN 2nd, Chang JH, MacEwan IJ, Wolden SL, Wang D, Yock TI, Aridgides PD. Outcomes following radiation therapy for embryonal tumor with multilayered rosettes (ETMR): results from the Pediatric Proton/Photon Consortium Registry (PPCR). J Neurooncol. 2025 Sep;174(2):369-380. doi: 10.1007/s11060-025-05065-2. Epub 2025 May 13. PMID 40358803